CLINICAL TRIAL: NCT00112164
Title: Prospective, Randomized Phase II Clinical Trial of Activated Protein C (Xigris) Versus Placebo for the Treatment of Acute Lung Injury
Brief Title: Activated Protein C to Treat Acute Lung Injuries
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Per recommendation of the NHLBI DSMB
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 175; P50HL074005 (NIH)
Record Dates: First submitted 2005-05-27; First posted 2005-05-30 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — drotrecogin alfa activated

INTERVENTIONS:
Drug: Xigris

SUMMARY:
The purpose of this study is to test the efficacy of activated Protein C (Xigris) for improving clinical outcomes in individuals with acute lung injury (ALI).

DETAILED DESCRIPTION:
BACKGROUND:

The hypothesis that procoagulant and inflammatory mechanisms may have a dual role in tissue injury was tested in the phase III clinical trial of recombinant Xigris for severe sepsis (Bernard, 2001). There was a significant reduction in mortality from 30% to 24% in patients treated with Xigris. However, there is no information on the effect of Xigris on patients with sepsis and co-existing ALI. Because Xigris is known to have both anti-coagulant and anti-inflammatory properties, it is plausible that it may be effective at treating patients with ALI from pulmonary and non-pulmonary infectious causes. There is also a good rationale for the hypothesis that Xigris may be effective at treating ALI from non-infectious causes. In experimental lung injury, from a non-infectious cause, such as hyperoxia or a like acid-lung injury, pro-coagulant mechanisms play a role in the pathogenesis of the ALI (Eitzman, 1996; Barazzone, 1996). Furthermore, research has shown that plasma-protein C deficiency occurs in almost all patients with ALI, and reduced Protein C levels are associated with a higher mortality and more non-pulmonary organ system dysfunction, even in patients with non-septic causes of ALI (Ware, 2003). Elevated levels of thrombomodulin, a product of endothelial injury, were measured in the plasma of all patients with ALI regardless of the clinical disorder associated with lung injury. The elevations of thrombomodulin were much higher in edema fluid than in plasma, suggesting that local activation and release of thrombomodulin had occurred, probably from both epithelial and endothelial sources from the lung, again supporting the hypothesis that a common pathway to lung injury may occur in both septic and non-septic causes of ALI. In addition, there is considerable evidence that the normal fibrinolytic mechanisms are impaired in the alveolar compartment in patients with ALI. Elevated levels of plasminogen-activator-inhbitor-1 (PAI-1) in the plasma of pulmonary edema fluid have a predictive value for identifying patients with ALI who are more likely to die than survive, regardless of the clinical risk factors that predisposes the development of ALI (Prabhakaran, 2003). Thus, this supports the rationale for testing Xigris as a treatment for patients with ALI, regardless of the clinical disorder associated with the cause of the lung injury. Since Xigris has both anti-coagulant and anti-inflammatory properties (Esmon, 2000; Grey, 1994), this treatment could reverse both the intravascular and the extravascular lung injuries and allow the lung epithelial and endothelial barriers to recover from a functional breakdown of both barriers. This study will evaluate the effects of the treatment of biochemical markers on alveolar epithelial injury.

DESIGN NARRATIVE:

Participants will be randomly assigned to receive either Xigris or saline placebo, to be administered continuously for 96 hours. Participants will be followed for 28 days, regardless of whether the drug is stopped for an adverse event, if the participant or physician decides to stop the drug, if the participant is discharged from the hospital with unassisted breathing, or until death.

ELIGIBILITY:
Inclusion Criteria:

* PaO2/FiO2 levels less than or equal to 300
* Bilateral infiltrates consistent with pulmonary edema on frontal chest radiograph
* Positive pressure ventilation through an endotracheal tube or tracheostomy
* No clinical evidence of left atrial hypertension that would explain the pulmonary infiltrates; if measured, pulmonary arterial wedge pressure less than or equal to 18 mm Hg

Exclusion Criteria:

* Family / patient refuses
* Patient / surrogate unavailable
* Attending refuses
* Age younger than 18 years
* Severe sepsis and Acute Physiology and Chronic Health Evaluation (APACHE) II scores greater than 25 within 48 hours of onset of severe sepsis
* Greater than 72 hours since all inclusion criteria are met
* Neuromuscular disease that impairs ability to ventilate without assistance, such as C5 or higher spinal cord injury, amyotrophic lateral sclerosis, Guillain-Barré syndrome, myasthenia gravis, or kyphoscoliosis
* Pregnant
* Severe chronic respiratory disease
* Weighs more than 160 kg
* Burns to more than 70% of total body surface area
* Cancer or other irreversible disease or condition for which 6-month mortality is estimated to be greater than 50%
* Bone marrow transplant in the 5 years prior to study entry
* Not committed to full support
* Severe chronic liver disease, as determined by a Child-Pugh Score of 11 to 15
* Diffuse alveolar hemorrhage from vasculitis
* Participation in another experimental medication study within 30 days of study entry
* Patients who have already received APC therapy
* Active internal bleeding
* Hemorrhagic or ischemic stroke within 3 months of study entry
* Intracranial or intraspinal surgery or severe head trauma within 2 months of study entry
* Trauma with an increased risk of life-threatening bleeding
* Presence of an epidural catheter
* Intracranial neoplasm mass lesion or evidence of cerebral herniation
* High risk of intracranial hemorrhage, as determined by 1 of the following: 1) intracranial or spinal pathology which places individuals at risk for intracranial hemorrhage (e.g., arterio-venous malformation or previous intracranial bleeding events, not including meningitis); 2) acute change in neurological status with focal neurological findings; 3) documented intracranial hypertension by lumbar puncture or imaging; or 4) seizures in which there is a clinical suspicion of intracranial hemorrhage
* Known bleeding diathesis
* Concurrent therapeutic heparin (greater than 14 units/kg/hr)
* Platelet count less than 30,000 x 106/L, even if the platelet count is increased after transfusions
* Prothrombin time greater than 3.0 INR
* Gastrointestinal bleeding within 6 weeks of study entry
* Concurrent need for systemic anticoagulation with therapeutic unfractionated heparin or low molecular weight heparin during the study drug infusion
* Concurrent administration of an anticoagulant (other than subcutaneous heparin for prophylaxis)
* Concurrent need for platelet glycoprotein Iib/IIIa antagonists or any other antiplatelet agents (patients taking aspirin or other antiplatelet agents at study entry are eligible if medication can be discontinued during study drug infusion)
* Surgery within 30 days of study entry and single organ failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2005-01; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Number of ventilator-free days (measured at Day 28)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Matthay, Study Chair — University of California, San Francisco
Locations (9):
- United States (9):
  - University of California San Francisco at Fresno, Fresno, California
  - University of Southern California, Los Angeles, California
  - San Francisco General Hospital, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Stanford University, Department of Pulmonary and Critical Care, Stanford, California
  - Yale School of Medicine, Section of Pulmonary & Critical Care Medicine, New Haven, Connecticut
  - Joseph M. Still Burn Center, Augusta, Georgia
  - Bay State Medical Center, Springfield, Massachusetts
  - Oregon Health Sciences University, Portland, Oregon

REFERENCES:
- [Background] Ware LB, Matthay MA. The acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1334-49. doi: 10.1056/NEJM200005043421806. No abstract available. PMID 10793167
- [Background] Bernard GR, Vincent JL, Laterre PF, LaRosa SP, Dhainaut JF, Lopez-Rodriguez A, Steingrub JS, Garber GE, Helterbrand JD, Ely EW, Fisher CJ Jr; Recombinant human protein C Worldwide Evaluation in Severe Sepsis (PROWESS) study group. Efficacy and safety of recombinant human activated protein C for severe sepsis. N Engl J Med. 2001 Mar 8;344(10):699-709. doi: 10.1056/NEJM200103083441001. PMID 11236773
- [Background] Nuckton TJ, Alonso JA, Kallet RH, Daniel BM, Pittet JF, Eisner MD, Matthay MA. Pulmonary dead-space fraction as a risk factor for death in the acute respiratory distress syndrome. N Engl J Med. 2002 Apr 25;346(17):1281-6. doi: 10.1056/NEJMoa012835. PMID 11973365
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Derived] Liu KD, Levitt J, Zhuo H, Kallet RH, Brady S, Steingrub J, Tidswell M, Siegel MD, Soto G, Peterson MW, Chesnutt MS, Phillips C, Weinacker A, Thompson BT, Eisner MD, Matthay MA. Randomized clinical trial of activated protein C for the treatment of acute lung injury. Am J Respir Crit Care Med. 2008 Sep 15;178(6):618-23. doi: 10.1164/rccm.200803-419OC. Epub 2008 Jun 19. PMID 18565951